CLINICAL TRIAL: NCT00064571
Title: Medialization Vs Reinnervation for Vocal Cord Paralysis
Brief Title: Surgery for Vocal Cord Paralysis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: U01DC004681 (NIH)
Record Dates: First submitted 2003-07-09; First posted 2003-07-10 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Unilateral Vocal Cord Paralysis
Keywords: unilateral vocal fold paralysis
MeSH Terms: conditions — Vocal Cord Paralysis

INTERVENTIONS:
Procedure: vocal fold medialization
Procedure: vocal fold reinnervation

SUMMARY:
Unilateral vocal fold paralysis (UVFP) is caused by injury to the nerve to the affected vocal fold. The injury to the vocal fold makes the affected person's voice sound "breathy". Voice therapy is usually tried first, and, if unsuccessful, surgical treatment is considered. The standard surgical treatment is called vocal fold medialization and aims to bring the injured cord to the midline. An alternative surgical treatment, vocal fold reinnervation, aims to bring a new nerve supply to the injured vocal fold. The reinnervation operation, which has some potential advantages over the medialization operation also requires several months for final results to be gained. The goal of this multicenter, randomized clinical trial is to see which of the two surgical treatments produces a better outcome.

In order to participate in this study patients with UVFP must meet all entry criteria and must be released from voice therapy by a speech-language pathologist. Information collected for the study (pre-surgery, and at 6 and 12 months after surgery) includes voice recordings, movies made of vocal fold function, airflow and pressure measurements of the voicebox, and an outcomes questionnaire.

DETAILED DESCRIPTION:
Unilateral vocal fold paralysis (UVFP) is caused by injury to the recurrent laryngeal nerve. Patients with UVFP may have significant impairment of vocal fold function, including a breathy paralytic dysphonia. There are several available approaches for the treatment of this condition. Vocal fold medialization is currently used by most otolaryngologists and is probably the standard of care for treating UVFP. An alternative approach is laryngeal reinnervation, which has a number of potential advantages over medialization but which requires several months before a final result is achieved. The primary goal of this multicenter, randomized clinical trial is to determine which approach produces a better outcome.

Patients with UVFP meeting all inclusion criteria and released from therapy by a speech-language pathologist will be randomized into either the medialization arm or the reinnervation arm. The data collection protocol consists of voice recordings, aerodynamic measurements, electroglottography, videostroboscopy, and a clinical outcomes questionnaire collected pre-treatment and at 6 and 12 months post-treatment.

ELIGIBILITY:
Inclusion criteria

* clinical diagnosis of unilateral vocal fold paralysis
* older than 18 years of age
* intact ansa cervicalis and recurrent laryngeal nerves
* life expectancy of greater than 2 years
* onset of the vocal fold paralysis within 2 years of the time of surgery
* no gelfoam injection for at least 4 months prior to initial data collection
* able to give informed consent
* willing and able to return for 6 and 12 month data collection sessions
* able and willing to perform questionnaire (by mail) 18 months after surgery

Exclusion criteria

* abnormal non-paralyzed fold
* other disorders affecting the larynx (voice box), such as multiple sclerosis, myasthenia gravis, spasmodic dysphonia, or essential voice tremor
* prior surgery to either vocal fold
* previous or planned irradiation of the voicebox

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-10; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Randal C Paniello, MD, Principal Investigator — Washington University School of Medicine
Locations (12):
- United States (12):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - UC-Irvine Medical Center, Irvine, California
  - George Washington University, Washington D.C., District of Columbia
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin